# **Mobile Mental Health Apps for Suicide Prevention**

NCT number: NCT04536935

**Document Date:** 12/22/2020

#### UNIVERSITY OF WASHINGTON

# Acceptability, Usability and Effectiveness of Mental Health Apps for Suicide Prevention in Essential Workers and the Unemployed during COVID-19

# **Randomized Trial Phase Consent Form**

The University of Washington is conducting a research study to learn about the acceptability, feasibility, usability, and effectiveness of mobile mental health apps for addressing risk factors associated with suicide risk in essential workers and unemployed individuals during COVID-19.

#### STUDY PROCEDURES

Thank you for answering our initial questions! If you agree to participate in this phase of the study, you will be randomly assigned to use one of 4 mobile mental health apps for 4 weeks. We'll ask you to complete a brief survey about your mood before we let you know which app you have been assigned to use. After completing those questions, we will ask you to download the app to your mobile device and interact with it for 4 weeks. We anticipate that answering these questions will take about 5 minutes. After completion of these questions, you will be paid \$1.

At the end of the 4 weeks, we will contact you through mTURK or Prolific to complete questions about your experience using the app and your mood, mental health, and well-being. We anticipate that answering these questions will take about 15 minutes. After completion of these questions, you will be paid \$4.

Only meaningful responses will be considered a completed survey. Meaningful responses are determined by successful completion of the entire survey, reasonable completion time, and passing quality checks. Quality checks are questions in the survey that anyone can answer correctly if thoughtfully reading the question. You must submit the HIT to receive compensation. Only submitted HITs with complete responses, reasonable response time, and passing quality checks will be accepted. If you submit a HIT for a survey response that does not meet these requirements, your HIT will be rejected. If you are not compensated, please contact the study team through the messaging system within mTURK or Prolific to receive a detailed explanation of why your data did not reach the standards.

Some of the questions that we ask may be uncomfortable to answer since we are asking some personal questions about your mood and mental health. You may refuse to answer any question at any time and continue with the study. The interview may result in fatigue; however, you may take breaks during the interview if you choose.

# **SOURCE OF FUNDING**

The University of Washington is receiving financial support from the National Institute of Mental Health.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **BENEFITS OF THE STUDY**

There will be no direct benefit to you from participating in the study, although you will receive information on mobile mental health apps that you may find helpful.

### **CONFIDENTIALITY OF RESEARCH INFORMATION**

The study team maintains the confidentiality of research information, meaning that no one other than the people working on the study will see your answers to the questions, unless required by law. We have a Certificate of Confidentiality from the federal National Institutes of Health. This helps us protect your privacy. The Certificate means that we do not have to give out information, documents, or samples that could identify you even if we are asked to by a court of law. We will use the Certificate to resist any demands for identifying information.

We can't use the Certificate to withhold your research information if you give your written consent to give it to an insurer, employer, or other person. Also, you or a member of your family can share information about yourself or your part in this research if you wish.

There are some limits to this protection. We will voluntarily provide the information to:

- a member of the federal government who needs it in order to audit or evaluate the research;
- individuals at the institution(s) conducting the research, the funding agency, and other groups involved in the research, if they need the information to make sure the research is being done correctly;
- the federal Food and Drug Administration (FDA), if required by the FDA;
- individuals who want to conduct secondary research if allowed by federal regulations and according to your consent for future research use as described in this form;
- local authorities, if we learn of child abuse, elder abuse, or the intent to harm yourself or others.

The Certificate expires when the NIH funding for this study ends. Currently this is April 30, 2022. Any data collected after expiration is not protected as described above. Data collected prior to expiration will continue to be protected.

# **USE OF INFORMATION**

The information and/or data that we obtain from you for this study might be used for future research. We will have no access to anything that might identify you so nothing identifiable would be shared. If we do so, that information and data may then be used for future research

# Approved 12/22/2020 UW IRB

studies or given to another investigator without getting additional permissions from you. It is also possible that in the future we may want to use or share study information that might identify you. If we do, an independent review board will decide whether or not we need to get additional permissions from you.

#### OTHER INFORMATION

There is no cost to you for participating in the study. However, downloading and using the mobile mental health application may count against your mobile data plan. You may change the settings on your phone to only use WiFi. The study will not provide any compensation or reimbursement for charges against your mobile plan.

Participation in research is voluntary and you may refuse or discontinue with no penalty. An alternate to participation is that mental health apps are available for you to seek out, download, and use even if you do not enroll in the study.

If you have questions about the research or think you have been harmed, you may contact the study team at (206) 744-1752 or <a href="mailto:uwcspar@uw.edu">uwcspar@uw.edu</a>. If you have questions about your rights as a subject, you can contact the UW Human Subjects Division at <a href="mailto:hsdinfo@uw.edu">hsdinfo@uw.edu</a>.

Because this is a research study, it is important that you know what is going to happen. Please answer these questions:

Being in the research study is voluntary. TRUE/FALSE

True: That's right! Being in this study is completely voluntary and you can stop at any time.

False: Good try! Actually, being in this study is voluntary and you can stop at any time.

I will be randomly assigned to use a mental health app for the next 4 weeks. I will not be able to choose which app I am asked to use. TRUE/FALSE

True: That's right! Neither you nor the study team gets to pick which app you use for the study. You are randomly assigned to an app – just like flipping a coin.

False: Almost! Neither you nor the study team gets to pick which app you use for the study. You are randomly assigned to an app – just like flipping a coin.

No one other than the people working on the study will see my answers to the questions, unless the study is being reviewed by individuals at UW, the funding agency, and other groups involved in the research if they need the information to make sure the research is being done correctly. TRUE/FALSE

True: That's right! We will keep all of your answers private, unless the study is being reviewed by individuals at UW, the funding agency, and other groups involved in the research if they need the information to make sure the research is being done correctly.

Approved 12/22/2020 UW IRB

False: Nice try! We actually do keep all of your answers private, unless the study is being reviewed by individuals at UW, the funding agency, and other groups involved in the research if they need the information to make sure the research is being done correctly.

| Thanks for answering our questions. Now is the time to let us know whether or not you would like to participate in the study. Please check one of the boxes below. | |
|---|---|
| | Yes, I agree to take part in this study. |
| | No, I do not want to take part in this study. |